CLINICAL TRIAL: NCT00545961
Title: Clinical Relevance of Middle Meatal Bacteriology During Acute Respiratory Infection in Children - Randomised, Double-Blinded Clinical Study
Brief Title: Middle Meatal Bacteriology During Acute Respiratory Infection in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oulu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Diary nr 41/2007
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Acute Respiratory Infection; Sinusitis
Keywords: respiratory infection; sinusitis; rhinosinusitis; children; middle meatal specimens; respiratory track bacteria; amoxicillin-clavulanate; pneumococci; haemophilus; moraxella
MeSH Terms: conditions — Sinusitis; Respiratory Tract Infections; Rhinosinusitis; Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo Ora-Plus (registered trademark) mixture with an strawberry sweetening agent to make the placebo mixture similar in appearance and taste to active drug
  Interventions: Drug: placebo
- 2 (Active Comparator): amoxicillin-clavulanate acid
  Interventions: Drug: amoxicillin clavulanate acid

INTERVENTIONS:
Drug: placebo — mixture, 0.28125 ml/kg twice a day for 7 days
  Other Names: Ora-Plus (registered trademark) mixture
  Arms: 1
Drug: amoxicillin clavulanate acid — mixture 0.28125 ml / kg twice a day for 7 days
  Other Names: Clavurion mixture (Orion Oy)
  Arms: 2

SUMMARY:
The purpose of this study is to find out whether the children with respiratory infection and the presence of pathogenic bacteria (S. pneumoniae, H. influenzae or M. catarrhalis) in the nasal middle meatus benefit from antimicrobial treatment.

DETAILED DESCRIPTION:
Acute sinusitis is one of the most common disease in children requiring antimicrobial treatment. The diagnosis and treatment outcomes of acute sinusitis are contradictory, and better diagnostic criteria are needed. In adults with acute maxillary sinusitis, bacterial culture results obtained from the nasal middle meatus are comparable to those obtained from sinus puncture and aspiration. In children, the presence of pathogenic bacteria (S. pneumoniae, H. influenzae or M. catarrhalis) in the nasal middle meatus during respiratory infection predicts longer duration of signs and symptoms of common cold.

In this randomized placebo-controlled study, the effect of the antimicrobial treatment (amoxicillin-clavulanate) is examined in children with pathogenic bacteria (S. pneumoniae, H. influenzae or M. catarrhalis) in the nasal middle meatus during respiratory infection. The duration of the symptoms and speed of recovery is recognized by daily symptom-diary, the results are compared between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory infection with nasal symptoms (nasal obstruction or discharge)
* seeking medical help from health centre for the respiratory symptoms
* pathogenic bacteria (S pneumoniae, H influenzae or M catarrhalis) identified from right or left nasal middle meatus in the endoscopically taken swab culture sampling taken by a study investigator (all microbiological analyses are done by the National Public Health Institute´s microbiological laboratory in Oulu)

Exclusion Criteria:

* otitis, tonsillitis or other disease requiring antimicrobial treatment
* respiratory infection within 4 weeks of screening
* antimicrobial treatment within 4 weeks of screening
* allergy to penicillin or amoxicillin

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2007-11; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Duration of continuous daily symptoms of the acute respiratory infection diagnosed at the study entry. | within the first 3 weeks after enrolment

SECONDARY OUTCOMES:
duration (days)and severity (grade mild, severe) of different symptoms (clear nasal discharge, coloured nasal discharge, nasal obstruction, cough, throat pain, ear ache, fever, headache, diarrhea) | within the first three weeks after enrolment
number of days the child is using the following symptomatic drugs (pain killers, nasal vasoconstrictors, nasal corticosteroids, asthma drugs, antihistamines) | within the first three weeks after the enrolment
number of days the child is not at school and that the parents are not at work | within the first three weeks after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jukka-Pekka Kuusiniemi, MD, Principal Investigator — Dept of Otolaryngology, Seinäjoki Central Hospital, Finland; Eeva Löfgren, MD, Principal Investigator — Dept of Otolaryngology, Kokkola Central Hospital, Finland; Anna Marttila, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Olli-Pekka Alho, professor, Study Director — Dept of Otolaryngology, University of Oulu, Finland; Aila Kristo, MD, Study Director — Dept of Otolaryngology, University of Oulu, Finland; Ulla Lantto, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland
Locations (3):
- Finland (3):
  - Keski-pohjanmaan keskussairaala, Kokkola
  - Oulu University Hospital, Oulu
  - Etelä-Pohjanmaan Keskussairaala, Seinäjoki